CLINICAL TRIAL: NCT00714168
Title: The Effect of a Stepped-care Approach to Long-term Weight Loss
Brief Title: Evaluating the Effectiveness of a Stepped-Care Approach to Long-Term Weight Loss (The Step-Up Study)
Acronym: Step-Up
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, John M. Jakicic, PhD, Professor and Chair, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 584; R01HL084400-04 (NIH); HL 084400
Record Dates: First submitted 2008-07-10; First posted 2008-07-14 (Estimated); Results first posted 2016-02-01 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2015-12

CONDITIONS: Obesity
Keywords: Weight Loss; Weight Control
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Participants will take part in a standard behavioral weight loss program.
  Interventions: Behavioral: Standard Behavioral Weight Loss Program
- 2 (Experimental): Participants will take part in a stepped-care weight loss program.
  Interventions: Behavioral: Stepped-Care Weight Loss Program

INTERVENTIONS:
Behavioral: Standard Behavioral Weight Loss Program — This program will include group sessions that will focus on modifying eating and physical activity behaviors to improve weight loss.
  Arms: 1
Behavioral: Stepped-Care Weight Loss Program — In this program, increases in the intensity of treatment will be based on participants' abilities to achieve predetermined weight loss goals. Participants will initially receive less contact with program staff. The intensity and/or frequency of contact will then increase at 12-week intervals, based on weight loss progress until a 10% weight loss is attained and maintained. The program will stay constant, unless weight loss drops below the 10% level.
  Arms: 2

SUMMARY:
The number of overweight and obese adults in the United States is increasing at a rapid rate. A "stepped-care" weight loss program, which at key times increases the frequency of contact between an individual trying to lose weight and the program staff, may be beneficial for achieving long-term weight loss. This study will compare a standard behavioral weight loss program with a "stepped-care" weight loss program in their abilities to help people who are overweight or obese to lose weight.

DETAILED DESCRIPTION:
Obesity can lead to many serious health conditions, including high blood pressure, diabetes, heart disease, and stroke. It is estimated that more than 65% of adults in the United States are overweight or obese, which is a significant increase over the past two to three decades. Although numerous studies have identified successful programs that help people achieve initial weight loss, few weight loss programs have shown promise for long-term success. Research has shown that a weight loss program in which there is continued contact between the program leader and the participant may improve long-term weight loss outcomes. In addition, a stepped-care approach to weight loss, in which contact between the participant and program leader increases when needed to achieve the next weight loss goal, may be beneficial. This study will examine whether a long-term weight loss program delivered in a stepped-care manner results in greater weight loss than does a standard behavioral weight loss program. Study researchers will also evaluate the cost effectiveness of both programs.

Participants in this 18-month study will be randomly assigned to either a standard behavioral weight loss program or a stepped-care weight loss program. Participants in the standard behavioral weight loss program will attend group meetings once a week for Months 1 to 6, every other week for Months 7 to 12, and once a month for Months 13 to 18. The group meetings will focus on modifying eating habits and physical activity behaviors to improve weight loss. Participants in the stepped-care weight loss program will take part in a combination of treatments, whose timing and intensity will depend on the participants' abilities to achieve predetermined weight loss goals. These treatments may include attending monthly group meetings, receiving weekly weight loss information in the mail, receiving telephone calls from study staff to discuss weight loss behaviors, taking part in individual sessions with study staff to discuss weight loss, and receiving meal replacements (e.g., Slim Fast shakes, meal bars). Participants who do not achieve their weight loss goals at select time points during the study will receive more individual attention from study staff. All participants will follow a diet that focuses on decreasing calories and fat. They will be instructed to follow a walking program 5 days a week and to keep a food and exercise diary. Participants will also have access to a Web site that will include a study calendar and information about how to change eating and exercise behaviors; the use of this Web site is optional.

Study visits will occur at baseline and Months 3, 6, 9, 12, 15, and 18. At each visit, participants' weight and height will be measured, and participants will complete questionnaires about their mood, general health, and exercise and diet habits. At baseline and Months 6, 12, and 18, participants will undergo measurements of blood pressure, fat, muscle, and waist and hip circumferences. Also at these times, physical fitness levels will be measured through a treadmill walking activity, during which an electrocardiogram (ECG) will record heart rate. For 7 consecutive days at baseline and Months 6, 12, and 18, participants will wear an activity monitor to measure physical activity levels.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 25.0 and 39.9 kg/m2

Exclusion Criteria:

* Reports losing more than 5% of current body weight in the 6 months before study entry
* Participated in a research project involving weight loss or physical activity in the 6 months before study entry
* Pregnant during the 6 months before study entry, currently breastfeeding, or planning to become pregnant in the 18 months after study entry
* Current treatment for any medical condition that could affect body weight (e.g., diabetes mellitus, cancer)
* History of heart attack or heart surgery, including bypass or angioplasty
* Currently taking medication that would affect heart rate or blood pressure responses to exercise (e.g., beta blockers)
* Currently taking medication that could affect metabolism or change body weight (e.g., synthroid)
* Currently being treated for psychological issues or has taken psychotropic medications in the 6 months before study entry

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 363 (Actual)
Dates: Start 2008-03; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John M. Jakicic, PhD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - University of North Carolina, Chapel Hill, North Carolina
  - University of Pittsburgh, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Creasy SA, Lang W, Tate DF, Davis KK, Jakicic JM. Pattern of Daily Steps is Associated with Weight Loss: Secondary Analysis from the Step-Up Randomized Trial. Obesity (Silver Spring). 2018 Jun;26(6):977-984. doi: 10.1002/oby.22171. Epub 2018 Apr 6. PMID 29633583
- [Derived] Davis KK, Tate DF, Lang W, Neiberg RH, Polzien K, Rickman AD, Erickson K, Jakicic JM. Racial Differences in Weight Loss Among Adults in a Behavioral Weight Loss Intervention: Role of Diet and Physical Activity. J Phys Act Health. 2015 Dec;12(12):1558-66. doi: 10.1123/jpah.2014-0243. Epub 2015 Mar 5. PMID 25742122
- [Derived] Jakicic JM, Tate DF, Lang W, Davis KK, Polzien K, Rickman AD, Erickson K, Neiberg RH, Finkelstein EA. Effect of a stepped-care intervention approach on weight loss in adults: a randomized clinical trial. JAMA. 2012 Jun 27;307(24):2617-26. doi: 10.1001/jama.2012.6866. PMID 22735431

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment included television and newspaper advertisements. Participants were enrolled between May 2008 and February 2010 at 2 clinical sites: 1) University of Pittsburgh, 2) University of North Carolina - Chapel Hill.
Pre-assignment Details: 433 individuals attended an orientation and provided written informed consent. Of these, 70 did not schedule a baseline assessment, failed to show for a baseline assessment, or were found to be ineligible after written consent was obtain. Thus, 363 were randomized to participate in this study.
Groups:
- Standard Behavioral Weight Loss Program: Participants will take part in a standard behavioral weight loss program.
  Standard Behavioral Weight Loss Program : This program will include group sessions that will focus on modifying eating and physical activity behaviors to improve weight loss.
- Stepped-Care Weight Loss Program: Participants will take part in a stepped-care weight loss program.
  Stepped-Care Weight Loss Program : In this program, increases in the intensity of treatment will be based on participants' abilities to achieve predetermined weight loss goals. Participants will initially receive less contact with program staff. The intensity and/or frequency of contact will then increase at 12-week intervals, based on weight loss progress until a 10% weight loss is attained and maintained. The program will stay constant, unless weight loss drops below the 10% level.
Period: Overall Study
Arm/Group | Standard Behavioral Weight Loss Program | Stepped-Care Weight Loss Program
Started | 165 | 198
Completed | 121 | 139
Not Completed | 44 | 59
Not completed — Pregnancy | 5 | 4
Not completed — Lost to Follow-up | 32 | 50
Not completed — Relocation | 4 | 3
Not completed — Non-study medical condition | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Behavioral Weight Loss Program | Stepped-Care Weight Loss Program | Total
Number analyzed (Participants) | 165 | 198 | 363
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 165 | 198 | 363
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.39 (9.22) | 42.04 (8.89) | 42.20 (9.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 136 | 164 | 300
  Male | 29 | 34 | 63
Region of Enrollment [Number; unit: participants]
  United States | 165 | 198 | 363

OUTCOME MEASURES:

1. Primary Outcome: Weight Loss
Description: Change in Weight from Baseline
Time Frame: Measured at Month 18
Population: We used an intention-to-treat analysis with all randomized subjects included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Arm/Group | Standard Behavioral Weight Loss Program | Stepped-Care Weight Loss Program
Number analyzed (Participants) | 165 | 198
kg | -8.1 [-9.4 to -6.9] | -6.9 [-8.0 to -5.8]

2. Secondary Outcome: Physical Activity
Description: Change in Physical Activity from Baseline
Time Frame: Measured at Month 18
Population: Intention-to-treat with all randomized subjects included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: kcal/week
Arm/Group | Standard Behavioral Weight Loss Program | Stepped-Care Weight Loss Program
Number analyzed (Participants) | 165 | 198
kcal/week | 700 [474 to 926] | 841 [627 to 1054]

3. Secondary Outcome: Energy Intake
Description: Change in Energy Intake from Baseline
Time Frame: Measured at Month 18
Population: Intention-to-treat with all randomized subjects analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: kcal/day
Arm/Group | Standard Behavioral Weight Loss Program | Stepped-Care Weight Loss Program
Number analyzed (Participants) | 165 | 198
kcal/day | -511 [-602 to -420] | -537 [-611 to -463]

4. Secondary Outcome: Cardiovascular Fitness
Description: Change in Minutes to achieve 85% of age-predicted maximal heart rate from Baseline
Time Frame: Measured at Month 18
Population: Intention-to-treat with all randomized subjects included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Standard Behavioral Weight Loss Program | Stepped-Care Weight Loss Program
Number analyzed (Participants) | 165 | 198
minutes | 2.7 [2.2 to 3.2] | 2.7 [2.3 to 3.1]

5. Secondary Outcome: Body Composition
Description: Change in Percent Body Fat from Baseline
Time Frame: Measured at Month 18
Population: Intention-to-treat with all randomized subjects included in the analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: percent body fat
Arm/Group | Standard Behavioral Weight Loss Program | Stepped-Care Weight Loss Program
Number analyzed (Participants) | 165 | 198
percent body fat | -5.6 [-6.4 to -4.8] | -5.0 [-5.7 to -4.3]

ADVERSE EVENTS:
Arm/Group | Standard Behavioral Weight Loss Program | Stepped-Care Weight Loss Program
Serious Adverse Events (participants affected / at risk) | 0/165 | 0/198
Other Adverse Events (participants affected / at risk) | 0/165 | 0/198

LIMITATIONS AND CAVEATS:
This study was not designed to test for weight loss equivalency between conditions. This study is unable to determined if an alternative intensity or frequency of intervention steps would be more or less effective for weight loss.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No